CLINICAL TRIAL: NCT02633423
Title: Expiratory Flow Limitation and Mechanical Ventilation During Cardiopulmonary Bypass in Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Elena Bignami, Professor, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EFLCCH
Record Dates: First submitted 2015-12-07; First posted 2015-12-17 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Mitral Regurgitation; Aortic Regurgitation
Keywords: Cardiopulmonary bypass; Mechanical ventilation; Expiratory Flow Limitation; Best PEEP
MeSH Terms: conditions — Mitral Valve Insufficiency; Aortic Valve Insufficiency | interventions — Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PEEP and CPAP (Experimental): Patients will be ventilated with positive end-expiratory pressure(PEEP) before and after cardiopulmonary bypass(CPB); during CPB continous positive airway pressure(CPAP) will be adopted.
  Interventions: Procedure: Use of PEEP before and after CPB; Procedure: Ventilation with CPAP during CPB
- ZEEP and CPAP (Experimental): Patients will be ventilated without PEEP(ZEEP) before and after cardiopulmonary bypass(CPB); during CPB continous positive airway pressure(CPAP) will be adopted.
  Interventions: Procedure: No use of PEEP before and after CPB(ZEEP); Procedure: Ventilation with CPAP during CPB
- PEEP and NO VM (Experimental): Patients will be ventilated with positive end-expiratory pressure(PEEP) before and after cardiopulmonary bypass(CPB); during CPB no mechanical ventilation will be adopted(no VM)
  Interventions: Procedure: Use of PEEP before and after CPB; Procedure: No ventilation during CPB
- ZEEP and NO VM (Placebo Comparator): Patients will be ventilated without PEEP(ZEEP) before and after cardiopulmonary bypass(CPB); during CPB no mechanical ventilation will be adopted(no VM)
  Interventions: Procedure: No use of PEEP before and after CPB(ZEEP); Procedure: No ventilation during CPB

INTERVENTIONS:
Procedure: Use of PEEP before and after CPB — PEEP will be set in order to reach an airway pressure of 5 cmH2O
  Arms: PEEP and CPAP; PEEP and NO VM
Procedure: No use of PEEP before and after CPB(ZEEP) — No PEEP will be used
  Arms: ZEEP and CPAP; ZEEP and NO VM
Procedure: Ventilation with CPAP during CPB — A continuous Positive Airway Pressure (CPAP) will be applied during CPB
  Arms: PEEP and CPAP; ZEEP and CPAP
Procedure: No ventilation during CPB — No ventilation will be provided during CPB. Patients will be deconnected from ventilator. Lungs will completely collapse.
  Arms: PEEP and NO VM; ZEEP and NO VM

SUMMARY:
During general anesthesia a reduction of Functional Residual Capacity (FRC) was observed. The reduction of FRC could imply that respiratory system closing capacity (CC) exceeds the FRC and leads to a phenomenon called expiratory flow limitation (EFL). Positive End-Expiratory Pressure (PEEP) test is a validated method to evaluate the presence of EFL during anesthesia. Aim of the study will be to asses if mechanical ventilation during CardioPulmonary Bypass (CPB) in cardiac surgery could reduce the incidence of EFL in the post-CPB period. Primary end-point will be the incidence of EFL, assessed by a PEEP test, performed at different time-points in operating room. Co-primary end-point will be shunt fraction, determined before and after surgery.

This will be a single center single-blind parallel group randomized controlled trial. Patients will be randomly assigned to four parallel arms with an allocation ratio 1:1:1:1, to receive one of four mechanical ventilation strategies during CPB.

1. Ventilation with a Positive End-Expiratory Pressure (PEEP) of 5 cmH2O before and after CPB; Continuous Positive Airway Pressure (CPAP) during CPB;
2. Ventilation without PEEP before and after CPB; CPAP during CPB;
3. Ventilation with a PEEP of 5 cmH2O before and after CPB; No use of mechanical ventilation during CPB
4. Ventilation without PEEP before and after CPB; No use of mechanical ventilation during CPB

DETAILED DESCRIPTION:
Introduction During general anesthesia a reduction of Functional Residual Capacity (FRC) was observed. The reduction of FRC could imply that respiratory system closing capacity (CC) exceeds the FRC and leads to a phenomenon called expiratory flow limitation (EFL). Several factors contribute to the EFL phenomenon during general anesthesia, including anesthesia induction by itself. High oxygen concentrations, muscle paralysis, supine positioning, increased extravascular water because of perioperative fluid therapy and inflammatory response also play a role in this picture.

Moreover cardiopulmonary bypass (CPB) with aortic cross-clamping, which is necessary for the majority of procedures in cardiac surgery, was associated with direct lung damage. Pulmonary atelectasis, apnea and ischemia during CPB and activation of proteolytic enzymes in the pulmonary circulation influence the incidence of postoperative pulmonary dysfunction after cardiac surgery.

Positive End-Expiratory Pressure (PEEP) test is a validated method to evaluate the presence of EFL during anesthesia. PEEP-test is a feasible and completely safe measure of the reduction of FRC in mechanically ventilated patients.

Aim of the study will be to assess if mechanical ventilation during CPB in cardiac surgery could reduce the incidence of EFL in the post-CPB period.

Primary End-point The primary endpoint will be a composite end-point of the incidence of Expiratory Flow Limitation after the weaning from CPB and post-operative pulmonary complications.

Secondary end-points

Secondary end-points will include:

* Readmission to the ICU;
* Need for re-intubation;
* Need for non-invasive ventilation;
* Duration of mechanical ventilation;
* Post-operative infections;
* Major adverse cardiac events;
* Length of the ICU and hospital stay;
* 30 days and 1 year mortality.

Materials and methods This will be a single center single-blind parallel group randomized controlled trial. Patients will be randomly assigned to four parallel arms with an allocation ratio 1:1:1:1, to receive one of four mechanical ventilation strategies during CPB. Patients that will match the following criteria at the preoperative evaluation will be recruited.

Randomization and masking Patient will be randomized according to a computer-generated list of casual numbers. Information about patient allocation will be kept in closed opaque envelopes and nobody will know patient allocation before randomization. Patients will be blind to allocation.

Ventilation protocol

Each patient will be randomized both about the ventilation management before and after CPB and about the management during CPB: a 2 by 2 trial design. Patients will be casually assigned to four groups:

Group A: patients will be ventilated with Positive End-Expiratory Pressure (PEEP) before and after cadiopulmonary bypass (CPB); during CPB, Continuous Positive Airway Pressure (CPAP) will be adopted.

Group B: patients will be ventilated without PEEP (ZEEP) before and after CPB; during CPB, CPAP will be adopted.

Group C: patients will be ventilated with PEEP before and after CPB; during CPB, no Mechanical Ventilation (No MV) will be adopted.

Group D: patients will be ventilated without PEEP (ZEEP) before and after CPB; during CPB, no MV will be adopted.

Patients will be randomized, immediately before surgery, to receive either a PEEP equal to the best PEEP, assessed with a PEEP test, immediately after the induction of anaesthesia or equal to zero. All patients will be furthermore randomized to receive either a CPAP equal to the best PEEP or a zero PEEP strategy (with deconnection from anaesthesia circuit) during CPB. The two randomizations will be independent each from other.

During CPB our goal will be to maintain PaO2 between 200 and 250 mmHg in order to avoid hyperoxia-induced lung injury; moreover, the hematocrit will be maintained above 24%.

During weaning from CPB we will perform a single alveolar RM. This RM will be performed manually by the anesthesiologist with a gas mixture of oxygen and air (with an inspired oxygen fraction lower than 80%) at the end of procedure. After CPB, this recruitment maneuver will be performed manually, in correspondence to the surgical de-airing procedure. Airway pressure will be kept at 40 cmH2O for at least 10 seconds.

Lung mechanics determination

Quasi-static compliance of respiratory system (Cqst,rs) will be calculated as:

Tidal volume / (end inspiratory plateau pressure - PEEPtot (ml/cmH2O) where PEEPtot is the end-expiratory pressure at period of no-flow. Measurement will be performed with an inspiratory pause of 60%.

Airway resistance (Rmin,rs) will be calculated as:

(Ppeak - P1) / V' where Ppeak is the peak inspiratory pressure, P1 is the airways pressure at the point of zero flow and V' is the inspiratory flow. Measurement will be performed with an inspiratory pause of 60%.

Lung mechanics will be determinated immediately after every PEEP test execution.

Dead space calculation

Dead space fraction calculation will be performed with the Enghoff modification of the Bohr equation:

Vd/Vt = (PaCO2-PECO2)/PaCO2

Where:

* Vd is the dead space
* Vt tidal volume
* PECO2 is pressure of mean expired CO2

Shunt fraction calculation

Shunt fraction will be determined before surgery and after surgery in operating room during general anesthesia, before patient discharge from operating room. Shunt fraction will be assessed as follows in all patients:

Qs/Qt = (PAO2 - PaO2)*0,0031 / C(a-v mixed)O2 + [(PAO2 - PaO2)*0,0031]

Where:

* PAO2 is oxygen alveolar concentration;
* PaO2 is oxygen arterial concentration;
* C(a-v mixed)O2 is arterovenous difference in oxygen concentration;
* 0,0031 is a conversion factor to volume percent for O2.

Measure will be performed while breathing 100% oxygen for 20 minutes, to achieve a complete hemoglobin saturation.

If a Pulmonary Artery Catheter (PAC) will be placed, according to clinical indications, shunt fraction will be calculated from the following formula:

Qs/Qt = CcO2-CaO2 / CcO2-Cv(mixed)O2 * 100

Where:

• CcO2 is pulmonary capillary blood O2 content, estimated with the following equation: CcO2 = (Hb * 1.34) + (0.0031 * PAO2);

* CaO2 is arterial oxygen content;
* Cv(mixed)O2 is oxygen content in blood samples obtained from the pulmonary artery;
* PAO2 is alveolar oxygen partial pressure. Blood samples will be collected from arterial catheter and pulmonary artery catheter, under a FiO2 of 100% in the same moment.

Furthermore Blood Gas Analyses (BGA) will be performed on arterial blood:

* after anesthesia induction;
* after sternotomy, together with heparinization;
* before sternosynthesis, together with protamine administration;
* before discharge from operating room.

Sample size calculation Sample size calculation was based on a 2 sided α error of 0.05 and a 80% power (β). On the basis of our experience, we anticipate that the 50% of patients with ventilation stop during CPB and no PEEP before and after CPB will reach the composite end-point of EFL after CPB and respiratory complications at 5 days, while only the 30% of the patients treated with an optimal. A sample size of 93 patients per group, 186 in total will be necessary to complete the trial. Including a drop-out fraction of 10%, we will enroll 51 patients per group, 204 in total.

Data collection and analysis Data will be collected on the appropriate Case Report Form (CRF). In particular anamnestic information will be collected, data about surgery and post-operative clinical data, in particular respiratory parameters. Data will be analyzed with a professional statistical software. Dichotomous variables will be compared with the two-tailed Chi square test, using the Yates correction when appropriate. Continuous variables will be compared by analysis of variance or the non-parametric Kruskal-Wallis test, when appropriate.

Informed consent and trial conduction Each patients will provide informed consent. All parts of this trial will be conducted according to the Good Clinical Practice (GCP) statement as well as Italian and international law on clinical research.

ELIGIBILITY:
Inclusion criteria:

* Elective cardiac surgery, with median sternotomy and two-lungs ventilation;
* Patients scheduled for mitral valve regurgitation and/or aortic valve regurgitation surgery, performed with CPB and aortic cross-clamping;
* Adult patients (age 18 or higher);
* Ability to provide informed consent.
* High risk for respiratory dysfunction, defined as 1 of: preoperative hypoxemia (arterial oxygen saturation < 92% in room air or arterial oxygen partial pressure < 60 mmHg at blood gas analysis or a PaO2/FiO2 ratio < 200 at basal blood gas analysis); preoperative obesity (BMI > 30); preoperative ejection fraction < 50%; preoperative NYHA class > II; age > 65 years.

Exclusion criteria:

* Non-elective cardiac surgery;
* Anticipated circulatory arrest, TAVI, Mitraclip;
* Patient's refusal;
* Pregnancy;
* Thoracotomic approach, with one lung ventilation;
* Previous pulmonary resection;
* Patients with acute kidney injury requiring dialysis;
* Patients with chronic kidney insufficiency (stage III or greater);
* Patients already intubated before arrival in operating theatre;
* Pneumonia in the previous 30 days.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2018-01-02 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of expiratory flow limitation in cardiac surgery | Immediately after weaning from cardiopulmonary bypass
Incidence of Postoperative pulmonary complications in cardiac surgery | From immediately after cardiac surgery until discharge from the hospital

SECONDARY OUTCOMES:
Duration of mechanical ventilation | Through study completion, an average of 24 hours after surgery
ICU length of stay | Through study completion, an average of 24 hours after surgery
Hospital length of stay | Through study completion, an average of 7 days after surgery
Re-admission to ICU | Through study completion, an average of 30 days after surgery
Need for reintubation | Through study completion, an average of 30 days after surgery
Need for non-invasive ventilation | Through study completion, an average of 30 days after surgery
Postoperative infections | Through study completion, an average of 30 days after surgery
Major adverse cardiac events | Through study completion, an average of 30 days after surgery
Incidence of mortality | Through study completion, 30 days and 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elena Bignami, MD, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, MI, Italy

REFERENCES:
- [Derived] Bignami E, Spadaro S, Saglietti F, Di Lullo A, Corte FD, Guarnieri M, de Simone G, Giambuzzi I, Zangrillo A, Volta CA. Positive end-expiratory pressure (PEEP) level to prevent expiratory flow limitation during cardiac surgery: study protocol for a randomized clinical trial (EFLcore study). Trials. 2018 Nov 26;19(1):654. doi: 10.1186/s13063-018-3046-0. PMID 30477541